CLINICAL TRIAL: NCT06924944
Title: Clinical Outcomes of Bilateral Clareon Vivity in Post-Refractive Patients
Status: Recruiting | Type: Observational
Sponsor: Utah Eye Centers (Other)
Responsible Party: Sponsor
Other Study IDs: UEC-101-001
Record Dates: First submitted 2025-01-22; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Correction Vision Surgery; Cataract Surgery
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Procedure: cataract surgery — cataract surgery treated with bilateral Clareon Vivity toric and non-toric IOL

SUMMARY:
Millions of people have undergone laser vision correction surgery and are motivated to continue with spectacle independence as they develop presbyopia (gradual loss of your eyes' ability to focus on nearby objects)and cataract. However, having a history of refractive surgery, poses challenges in the selection of the IOLs and can lead to visual outcomes that are unpredictable. Data from an international registry and single prospective study show that Vivity IOL provided effective distance, intermediate and near vision in eyes with previous LASIK with minimal effects on day vision associated with the surgery. The purpose of this study is to evaluate the clinical outcomes of post-myopic refractive surgery patients implanted with the Clareon Vivity/Vivity Toric lenses

ELIGIBILITY:
Inclusion Criteria:

* o Bilateral age-related visually significant cataracts in otherwise healthy eyes, undergoing uncomplicated bilateral sequential Clareon Vivity IOLs

  * Prior history of uncomplicated post-refractive myopic surgery (LASIK/PRK) with up to 1 enhancement treatment
  * Potential acuity measured post-operatively 20/25 or better in both eyes
  * Patients with regular astigmatism that can be managed with T3 toric lens or arcuate incision

Exclusion Criteria:

* o Ocular or systemic comorbidities that may alter or reduce visual acuity and contrast sensitivity such as severe dry eye/ocular surface disease, glaucoma, macular degeneration, retinopathy, neuro-ophthalmic diseases, etc.

  * Prior ocular surgeries other than uncomplicated corneal refractive surgery and excluding RK
  * Patients with irregular astigmatism/topography (to rule out signs of potential ectasia), corneal dystrophies, and pupil abnormalities
  * Total HOA cutoff of ≤0.5, coma ≤0.3
  * RLE patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult subjects with bilateral age-related cataract patients with history of myopic refractive surgery (LASIK/PRK)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Binocular photopic uncorrected distance VA (at 3 months) | at 3 months

SECONDARY OUTCOMES:
• Binocular photopic uncorrected VA at intermediate (66cm) and near (40cm) | at 3 months

OTHER OUTCOMES:
Monocular uncorrected distance, intermediate, and near VA | at 3 months
Monocular and binocular best distance corrected distance, intermediate, and near VA | at 3 months
Binocular photopic low contrast distance corrected VA | at 3 months
Mean refractive spherical equivalent (MRSE) for dominant and non-dominant eye | at 3 months
Mean difference of MRSE between dominant and non-dominant eye | at 3 months
% of eyes with absolute prediction error less than or equal to 0.5D | at 3 months
Visual disturbances via QUVID questionnaire | at 3 months
Potential association between HOA (SA and coma) and monocular DCVAs | at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Utah Eye Centers, Ogden, Utah, United States

IPD SHARING:
Plan to Share IPD: No